CLINICAL TRIAL: NCT04027673
Title: TMW-Early Childhood Educator Program
Brief Title: Thirty Million Words-Early Childhood Educator (TMW-ECE)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Chicago (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: IRB19-0602
Record Dates: First submitted 2019-07-11; First posted 2019-07-22 (Actual); Last update posted 2020-04-09 (Actual); Status verified 2020-04

CONDITIONS: Language Development

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment (Experimental): Participants in the treatment group complete interactive modules. They will be asked to complete one module per week, for a total of eight weeks.
  Interventions: Behavioral: TMW ECE Curriculum
- Control (No Intervention): Participants in the control group will have no active study requirements for the eight weeks following Survey Session 1.

INTERVENTIONS:
Behavioral: TMW ECE Curriculum — The TMW-ECE program will constitute the treatment arm of the study (Cohort A) which will complete the multi-media online professional development course beginning Summer 2019.
  Arms: Treatment

SUMMARY:
The purpose of the proposed study is to determine the efficacy of an eight-module interactive, online multi-media professional development course on our target population: individuals over the age of 18, who have no more than a bachelor's degree, and are employed as early childhood educators of children between the ages of 0 and 3. Outcomes of interest include changing caregiver knowledge and beliefs about child development, and encouraging the use of strategies provided to strengthen early learning environments. The investigators will also measure how participants interact with the online course in order to determine which features help and hinder the online professional development process.

The investigators hypothesize that the TMW-ECE intervention will be effective in improving educator beliefs and knowledge of their role in children's foundational brain development, and increasing the frequency of behaviors that are known to support children's language and cognitive development among our target population.

DETAILED DESCRIPTION:
The intervention modules are experimental. The modules will be completed by subjects online using their own computer and internet connection.

TMW will send email reminders to participants whose participation has lapsed for more than 3 weeks (no activity in the learning management system (LMS) during that time).

Phase 1: Pre-Intervention Participant completes a demographics survey on RedCap to determine eligibility based on the exclusion criteria listed below. If they are eligible and desire to participate, they will complete the informed consent process online prior to beginning the intervention.

Participants will be randomized into either the treatment or control group after providing their consent. All participants will be notified via email with detailed instructions on how to complete the study measures online and, if treatment group, how to view the modules.

Survey Session 1: Participant completes the following surveys online: Survey of Parent/Provider Expectations and Knowledge (SPEAK), Course Content Survey, and Theories of Intelligence (TOI).

Phase 2: Intervention Participants in the treatment group complete interactive modules. They will be asked to complete one module per week, for a total of eight weeks.

Participants in the control group will have no active study requirements for the eight weeks following Survey Session 1.

Phase 3: Post-Intervention Upon completion of Module 8, participants in the treatment group will be invited by email to complete Survey Session 2, which includes the following surveys: SPEAK,Theories of Intelligence (TOI) survey, Course Content Knowledge, and the qualitative Course Experience survey.

Participants in the control group will be invited to complete Survey Session 2 exactly eight weeks after they complete Survey Session 1, which corresponds to how long the investigators anticipate treatment group participants needing to complete the 8 modules. This Survey Session will include the same surveys as the treatment group: SPEAK, Theories of Intelligence (TOI) survey, Course Content Knowledge, and a qualitative Course Experience survey on their most recent professional development.

All participants in both experimental groups will be invited by email to complete Survey Session 3 exactly 12 weeks after the completion of Survey Session 2. Surveys include: SPEAK, Course Content Knowledge, and Theories of Intelligence (TOI) survey.

At the conclusion of the study, participants in the treatment group may be asked to participate in a phone interview about their experience with the program, their opinions on the curriculum, and how they interact with the children in their care. This interview will be conducted with a trained member of the research team. The investigators hope to interview all treatment group participants but are limited in human capacity to complete the phone interviews for our expected recruitment goals. The investigators will ask as many treatment group members to participate in the phone interview but will start with the most engaged participants and those who enrolled first.

ELIGIBILITY:
Exclusion Criteria:

* Educators who report having a higher level of education (above a bachelor's degree, including any graduate school coursework).
* Educators who do not work with children ages 0-3 as their primary age group.
* Educators who are under the age of 18.
* Educators who do not have access to a computer or tablet with access to the internet.
* Anyone not employed by a childcare program (either home or center-based).
* Anyone whose role within a childcare setting is not that of an educator (primary teacher or assistant teacher)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 432 (Actual)
Dates: Start 2019-06-03 (Actual); Primary Completion 2020-03-30 (Actual); Study Completion 2020-03-30 (Actual)

PRIMARY OUTCOMES:
Survey of Parent/Provider Expectations and Knowledge (SPEAK) | 6 months
  Provider knowledge of child language development
Course Content Knowledge | 6 months
  This survey includes questions specific to the course content conveyed in the professional development modules. True/false, and multiple-choice questions will measure participants' uptake of course material.
Tool to Measure Parenting Self Efficacy (TOPSE) | 6 months
  The TOPSE measures parents attitudes and beliefs about their parenting style and behaviors. In this study, it is administered only to participants who identified as having a child living in the home

SECONDARY OUTCOMES:
Experience survey | 3 months
  This survey asks about providers' experiences with the online professional development program format, including ease of use, opinions about the quality of the curriculum, suggestions for how the program can be improved in the future, and how providers have used what they learned in the curriculum in their own classroom.

CONTACTS AND LOCATIONS:
Overall Officials: Dana Suskind, MD, Principal Investigator — University of Chicago; Kristin Leffel, AB, Study Chair — University of Chicago
Locations (1):
- University of Chicago, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No
Descriptive IPD will not be shared

REFERENCES:
- [Background] Mashburn AJ, Pianta RC, Hamre BK, Downer JT, Barbarin OA, Bryant D, Burchinal M, Early DM, Howes C. Measures of classroom quality in prekindergarten and children's development of academic, language, and social skills. Child Dev. 2008 May-Jun;79(3):732-49. doi: 10.1111/j.1467-8624.2008.01154.x. PMID 18489424
- See also: Click here for more information about the Thirty Million Words — http://tmwcenter.uchicago.edu

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-07-19): https://cdn.clinicaltrials.gov/large-docs/73/NCT04027673/Prot_SAP_001.pdf